CLINICAL TRIAL: NCT00406289
Title: Phase I Trial of Adaptive 18F-FDG-PET Biological Intensity-modulated Radiotherapy (BG-IMRT) With Patients With Head and Neck Tumor
Brief Title: Trial of Adaptive 18F-FDG-PET Biological Intensity-modulated Radiotherapy (BG-IMRT) in Patients With Head and Neck Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Wilfried De Neve, University Hospital Ghent
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/391
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Head and Neck Tumor
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: 18F-FDG-PET radiotherapy

SUMMARY:
This study will evaluate the feasibility of higher and prolonged dose escalation concentrated in the intra-tumoral regions which are FDG-avid after two weeks of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck tumor
* Aged > 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Tumor recurrences

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be